CLINICAL TRIAL: NCT03069768
Title: Stage Ib Trial of mSMART With Varenicline
Acronym: mSMART-v
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to obtain varenicline to provide to participants
Sponsor: Duke University (Other)
Collaborators: Intelligent Automation, Inc. (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00080336; 271201400069C-0-0-1 (NIH)
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Nicotine Dependence
Keywords: Nicotine addiction; Cigarette smoking; Smoking cessation; Quit smoking
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mSMART (Experimental): Smokers in this group will have the mSMART application installed on their smartphones. The mSMART application will provide information about varenicline (Chantix) and reminders when it's time to take the medication.
  Interventions: Device: mSMART; Drug: Chantix
- Control (Active Comparator): Smokers in this group will not be given the mSMART application.
  Interventions: Drug: Chantix

INTERVENTIONS:
Device: mSMART — A smartphone application that targets medication adherence in substance users, providing information and reminders and tracking medication usage and factors interfering with adherence.
  Other Names: mSMART app; mSMART Smartphone Application
  Arms: mSMART
Drug: Chantix — For the first 3 days smokers in this group will receive treatment with Chantix at a dose of 0.5 mg once per day followed by 0.5 mg twice a day for the remaining 4 days of that week. Subsequently, the dose will be 1 mg twice per day, and will remain at that dose for the remainder of the 12-week active treatment duration.
  Other Names: Varenicline

SUMMARY:
The primary aim of this study is to conduct a 60-patient feasibility, acceptability, and preliminary efficacy study of mSMART (Mobile App based Personalized Solutions and Tools for Medication Adherence of Rx Pill), a smartphone application ("app") for improving medication adherence among substance users. The investigators will compare 2 groups of cigarette smokers undergoing a quit attempt with varenicline (Chantix): a) an experimental group using the mSMART app on their smartphone and a MEMS Cap (Medication Event Monitoring System, a smart pillbox that will a record a date and time-stamped medication event whenever pill box is opened and closed, and thus allow for primary measurement of medication adherence) and b) a control group using the MEMS Cap and mobile web-based surveys on their smartphone.

DETAILED DESCRIPTION:
Poor medication adherence (a) results in poorer treatment outcome and (b) accounts for $100 to $290 billion in U.S. healthcare costs annually. Therefore, interventions that target medication adherence are increasingly crucial for patient care and cost-effectiveness. Mobile technologies such as smartphones are increasingly ubiquitous and affordable in the U.S., and can be integrated to augment medication adherence. mSMART is a smartphone application that targets medication adherence in substance users. The study team has developed and assessed mSMART in a Stage Ia trial among 9 non-treatment seeking cigarette smokers. mSMART provides psychoeducation about medication (e.g., dosage, benefits, side-effects), assessment of medication compliance and characteristics associated with substance use, provides reminders to take medications, and conducts real-time medication event feedback intervention. The aim of the current study is to extend findings from the Stage Ia trial assessing preliminary feasibility and acceptability of mSMART for cigarette smokers. In the proposed study, the investigators will conduct a Stage Ib for the continued development of mSMART in an occupational wellness setting. This will also include a study of the feasibility, acceptability, and preliminary efficacy of mSMART for treatment seeking cigarette smokers undergoing a quit attempt. A sample of 60 cigarette smokers will be given varenicline (Chantix) and randomized to either a control condition (i.e., use of MEMS Cap, a smart pillbox that records instances that the pill bottle is opened) or treatment condition (i.e., use of MEMS Cap and mSMART) over a 12 week treatment period. The primary hypothesis is that the treatment group will achieve higher levels of medication adherence assessed via MEMS Cap. The secondary hypothesis is that the treatment group will also yield lower levels of salivary cotinine at week 12 assessment, indicating higher rates of smoking abstinence relative to the control group. Findings from the current study will inform the continued development of mSMART as an intervention to enhance substance use treatment outcome, including other forms of substance use besides cigarette smoking.

ELIGIBILITY:
Inclusion Criteria:

* Interested in taking varenicline (Chantix) with the intention to quit smoking in the next 3 months
* Has an Android smartphone (using v5.x.x or lollipop) or Apple smartphone (iPhone) Operating System (iOS) (using v6.0)
* 18-65 years of age

Exclusion Criteria:

* Unwillingness to be randomized to either treatment condition
* Subjects who have currently been taking varenicline for more than 15 days
* Currently pregnant or plan on becoming pregnant (females only)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Adherence to smoking cessation medication as assessed via Medication Event Monitoring System (MEMS) | Week 12
  The MEMS Cap, placed on the subject's medication bottle, will document the number of times the bottle is opened per day, totalled at the end of study
Acceptability of mSMART based on responses to an exit interview | Week 12
  Acceptability of mSMART will be based on responses to an exit interview at the end of the study (Visit 2). Questionnaire asks for agreement with statements relating to acceptability of the app. Response options will be quantified on a Likert scale (1 = not at all, 2 = somewhat, 3 = moderately, 4 = extremely). Example question: What was your overall satisfaction with mSMART?
Feasibility of mSMART based on frequency of participant use of the app | Week 12
  Feasibility of mSMART will be based on frequency of participant use of the app, totalled at the end of the study.

SECONDARY OUTCOMES:
Adherence to smoking cessation medication indicated by smoking abstinence | Week 12
  Adherence to smoking cessation medication will be evaluated by assessing a biochemical (salivary) measure of participant's cotinine level at the end of the 12 week intervention period which will assess smoking abstinence.
Adherence to smoking cessation medication indicated by mSMART medication event data | Week 12
  Adherence to smoking cessation medication analyzed using mSMART's medication event data from use of Medication Aide widget (a component of mSMART involving a smartphone camera-based medication identification and identification-based medication event technology developed by Intelligent Automation, Inc.) in the experimental group.

CONTACTS AND LOCATIONS:
Overall Officials: F. Joseph McClernon, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke Health Behavior Neuroscience Research Lab, Durham, North Carolina, United States